CLINICAL TRIAL: NCT04865146
Title: A Multicenter, Post Market, Clinical Follow-Up Study to Evaluate the Safety and Effectiveness of TRIGEN™ INTERTAN™ Intertrochanteric Antegrade Nails (10S Models) for the Treatment of Femoral Fracture in Chinese Subjects
Brief Title: A Study to Evaluate the Safety and Effectiveness of TRIGEN™ INTERTAN™ (10S Models)
Status: Withdrawn | Type: Observational
Why Stopped: Change on clinical and marketing strategy for intramedullary devices
Sponsor: Smith & Nephew Medical (Shanghai) Ltd (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: InterTan.2019.13
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Femoral Fractures; Hip Fractures
Keywords: femoral fractures; Nails; TRIGEN; INTERTAN
MeSH Terms: conditions — Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- TRIGEN™ INTERTAN™: Confirmed femoral fracture subjects who are scheduled for repair using INTERTAN 10S Nail
  Interventions: Device: TRIGEN™ INTERTAN™

INTERVENTIONS:
Device: TRIGEN™ INTERTAN™ — Femoral fracture treated with INTERTAN 10S Nail

SUMMARY:
This is a post-market study to evaluate the revision rate of femoral fractures, treated with INTERTAN 10S Nails at one-year post-operation. The study will enroll Approximately 180 subjects with femoral fractures, Approximately 7 sites are involved. The study duration will be Approximately 36 months (6 months start-up, 1 year enrollment, 1 year follow-up, 6 months closeout/study report).

DETAILED DESCRIPTION:
Background:

The INTERTAN nail was designed to improve upon existing intramedullary nail systems. INTERTAN nails utilize two interlocking screws, thereby improving controlled intertochanteric fracture compression and post-surgical stability.

Purpose:

Evaluate the revision rate of femoral fractures, treated with INTERTAN 10S Nails at one-year post-operation

Objectives:

* Primary Objective: To evaluate the revision rate for any reason of femoral fractures, treated with INTERTAN 10S Nails at one year post-operation
* Secondary Objective: To generate safety and effectiveness evidence for INTERTAN 10S Nails via the collection of functional outcomes, quality of life, and safety data

Research participants / locations:

The study will enroll Approximately 180 subjects with femoral fractures, Approximately 7 sites in China are involved.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who sign the informed consent form (ICF) voluntarily.
* Subjects who have a femoral fracture and are scheduled for repair using an INTERTAN 10S Nail.
* Male or female subjects aged 18 years or older, with mature bone development at time of implantation.
* Subjects who agree to follow all study visits and procedures.

Exclusion Criteria:

* Subjects with known hypersensitivity to the device or implant materials.
* Subjects in which use of the device would cross open epiphyseal plate(s).
* Subjects with complex intertrochanteric and femoral neck fractures.
* Subjects with an existing condition that predisposes them to a poor outcome, such as blood supply limitations, insufficient bone quality or quantity, obliterated medullary canal, previous infections or other conditions which tend to retard healing.
* Subjects not suitable for operation due to obvious local or systemic infection.
* Subjects who are unable to tolerate anesthesia and surgery due to cardiopulmonary failure or other serious diseases.
* Subjects with a congenital or acquired bony deformity.
* Subjects with Body Mass Index (BMI) of ≥ 35.
* Subjects with hypovolemia, hypothermia, or coagulopathy.
* Subject is immunosuppressed, has an autoimmune disorder or an immunosuppressive disorder. For examples, subjects are on immunosuppressive therapy (cortisol at large dose, cytotoxic drugs, antilymphocytic serum or irradiation at large doses) or has acquired immunodeficiency syndrome (AIDS).
* Subjects with any existing hardware that would preclude the use of the nail.
* Subjects with mental or emotional conditions or any other clinical conditions that, in the opinion of the Investigator, would preclude cooperation and compliance with the rehabilitation regimen.
* Subjects with medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* Subject is a woman who is pregnant or lactating, or intends to become pregnant during the course of the study follow-up.
* Subjects who have participated in any other clinical trial within 3 months of Screening.
* Subjects who have participated previously in this clinical study and were withdrawn for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who plan to be treated using TRIGEN™ INTERTAN™ (10S)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The Revision Rate | 1 year
  To evaluate the revision rate for any reason of femoral fractures, treated with INTERTAN 10S Nails at one year post-operation.

SECONDARY OUTCOMES:
Intraoperative Complications | Intraoperative
  Documentation of any complications related to the implantation of the device. Potential complications of this type of surgery include, but are not limited to, those listed below.
  * Loosening, bending, cracking or fracture of the implant components
  * Limb shortening or loss of anatomical position, accompanied with bone nonunion or with rotation or angulated malunion
  * Infections, both deep and superficial
  * Irritational injury of soft tissues, including impingement syndrome
  * Supracondylar fractures from retrograde nailing
  * Macrophage and foreign body reactions adjacent to implants
Radiographic Assessment | Pre-operative, 6 weeks, 3 months, 6 months, & 1 year
  Full-length standing radiographs, standard anteroposterior (AP), and lateral radiographs of lower extremities taken prior to surgery and at all follow-up time points to identify the presence of bone healing result, normal fracture healing and disturbed fracture healing.
Time to Union | Through study completion, approximately 1 year
  To evaluate the bone healing during each visit by achieving radiographic union.
Harris Hip Score (HHS) | 6 weeks, 3 months, 6 months, & 1 year
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worst) to 100 (best).
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Pre-operative, 6 weeks, 3 months, 6 months, & 1 year
  The EQ-5D-5L is a standardized instrument for use as a measurement of health outcome. It consists of a descriptive system with 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), which are each assigned five levels (no problems, slight problems, moderate problems, severe problems and extreme problems), as well as, a Visual Analogue Scale (VAS) where subjects indicate a numerical value from 1-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state.
  The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the dimensions. This decision results in a 1- digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Time to Return to Full Weight-Bearing | Post-operatively through study completion, approximately 12 months
  To evaluate the bone healing during each visit by achieving return to full weight-bearing.
Length of Stay | During hospitalization
  Length of stay in days participant spends in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqiang Sun, Principal Investigator — Shanghai 6th People's Hospital
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tang Shan 2rd Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Peking University Third Hospital, Beijing
  - Shanghai 6th People Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No